CLINICAL TRIAL: NCT03317873
Title: The Effect of Genetic Variation in TMPRSS6 Gene (SNP rs855791) on Oral Iron Absorption: an Iron Stable Isotope Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TMPRSS6_Fe
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Iron Metabolism Disorders
MeSH Terms: conditions — Iron Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wild type AA (CC) (Experimental): All participants with the wild type genotype AA (CC) will be allocated to this group
  Interventions: Dietary Supplement: Testmeal A; Dietary Supplement: Testmeal B
- mutation VV (TT) (Experimental): All participants with the mutation genotype VV (TT) will be allocated to this group
  Interventions: Dietary Supplement: Testmeal A; Dietary Supplement: Testmeal B

INTERVENTIONS:
Dietary Supplement: Testmeal A — The tesmeal A is is plain rice, with a seaweed sauce, fortified with labelled iron as stable iron isotope as ferrous sulfate
Dietary Supplement: Testmeal B — The tesmeal B is plain rice, with a seaweed sauce, fortified with labelled iron as stable iron isotope as ferrous sulfate

SUMMARY:
Iron deficiency is considered the most common nutritional deficiency worldwide and affects children and women in both non-industrialized as well as industrialized countries. The main regulatory molecule of iron metabolism is hepcidin, a hormone produced in the liver that regulates intestinal iron absorption, placental transport, recycling of iron by macrophages and release from stores. The expression of hepcidin is regulated by many mediators, one of which is Matriptase-2 - a transmembrane protease. Complete loss of function leads to the rare disease iron-refractory iron deficiency anemia (IRIDA). Matriptase-2 is encoded by the gene TMPRSS6 and the single nucleotide polymorphism (SNP) rs855791 causes a non-synonymous substitution (V736A) that reduces the activity of the protease to inhibit hepcidin transcription. Genome wide association studies have identified the TMPRSS6 SNP rs855791 has a strong association with red blood cell and iron parameters in the general population.

The objectives of the study is to measure oral iron absorption and systemic iron utilization into red blood cells (RBC) using oral isotopic labels in subjects homozygotes for common variants of the TMPRSS6 gene with the SNP rs855791 (A736V); AA vs. VV subjects.

The aim is to conduct an iron absorption study in 80 Taiwanese women of reproductive age, non-pregnant, non-anemic, investigating the effect of the genetic variants of the SNP rs855791. The participants will be split in two groups of equal size; wild type AA vs. mutation VV. Iron absorption and systemic utilization will be assessed by two test meals containing stable isotopes of iron.The primary outcome of the trial is the oral iron absorption from a test meal as compared between the two genotypes AA vs. VV. Secondary outcomes are the comparison iron status markers between the two genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects homozygotous for the for AA (CC), or VV (TT) variant of the SNP rs855791 of the TMPRSS6 gene.
* Females 20 - 45 years of age (premenopausal status)
* obtained informed consent
* regular menstrual cycle, ± 2 days

Exclusion Criteria:

* Pregnancy or lactating (assessed by pregnancy test and self-declaration, respectively)
* Anemia defined as Hb < 120 g/L
* Plasma ferritin < 30 µg/l, or > 120 µg/l
* C-reactive Protein > 5 mg/l
* Body weight > 65 kg
* Body mass index (BMI) 18.5 - 25
* Diagnosed metabolic or gastrointestinal disorders, eating disorders or food allergy to the ingredients of the test meal.
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 6 months, prior the first study day.
* Subjects who cannot be expected to comply with study protocol (e.g. non-residents).
* Use of long-term medication during the study
* Subjects that will take part of another clinical study at the same time or had within the last 30 days before the first study day
* Intake of mineral/vitamin supplements 2 weeks before the first study day and during the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron in blood will be measured after the administration of test meal including iron isotopes.

SECONDARY OUTCOMES:
hepcidin | baseline
  fasting concentrations of plasma hepcidin in AA and VV variants of SNP rs855791
iron status | baseline
  The difference in fasting concentrations of serum iron, transferrin saturation, serum ferritin, hemoglobin, erythrocyte volume in AA and VV variants of SNP rs855791

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung-Chang Gun Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Buerkli S, Pei SN, Hsiao SC, Lee CT, Zeder C, Zimmermann MB, Moretti D. The <em>TMPRSS6</em> variant (SNP rs855791) affects iron metabolism and oral iron absorption - a stable iron isotope study in Taiwanese women. Haematologica. 2021 Nov 1;106(11):2897-2905. doi: 10.3324/haematol.2020.264556. PMID 33054130